CLINICAL TRIAL: NCT02501564
Title: Randomized, Double-blind and Placebo-controlled Evaluation of Efficacy and Safety of Naproxen Sodium and Codeine Phosphate Combination in Osteoarthritis
Brief Title: Evaluation of NaproxenSodium and CodeinePhosphate Combination in Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Principal Investigator, KAYA AKAN, MD, Associate Professor, Associate Professor of Orthopedics and Traumatology, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAPCOD2013
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; NAPROXEN SODIUM
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen Sodium Codeine (Experimental): One tablet twice a day
  Interventions: Drug: Naproxen Sodium Codeine
- Placebo (Placebo Comparator): One tablet twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium Codeine — One tablet twice a day
  Other Names: Apranax Plus
  Arms: Naproxen Sodium Codeine
Drug: Placebo — One tablet twice a day
  Arms: Placebo

SUMMARY:
Osteoarthritis (OA) pain treatment has limitations in terms of serious adverse effects and low efficacy. The investigators aimed to evaluate efficacy and safety of naproxen sodium/codeine phosphate combination in these patients.

DETAILED DESCRIPTION:
In this prospective, randomized, double blind, placebo controlled clinical trial, 135 patients with osteoarthritis, who were 40-65 years; applied to institution's orthopaedics outpatient clinic; had grade 1, 2, or 3 primary osteoarthritis diagnosed in last 1 year; and had Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score≥40, and Visual Analogue Scale score≥40,were enrolled. Subjects were randomized (1:1) to placebo (n= 67) or combination (n= 68) arms, in which 550 mg naproxen sodium/30mg codeine phosphate was given orally twice a day for 7 days. Rescue medicine was 500 mg paracetamol (max= 6 tablets/day). Demographic characteristics, medical history, adverse events, VAS and WOMAC scores were collected in study visits performed within 10days.The study was approved by local institutional ethics committee and written informed consents were obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of primary osteoarthritis (knee and hip) in the recent year according to criteria of American College of Rheumatology (ACR)
* Grade 1, 2 or 3 osteoarthritis patients
* Patients 40 to 65 years of age
* Patients with WOMAC score ≥ 40
* Patients with VAS score ≥ 40
* Patients who signed the consent form

Exclusion Criteria:

* Grade 4 osteoarthritis patients / Pregnant or breastfeeding mothers
* Patients with known allergic reaction or intolerance to NSAIDs (nonsteroidal antiinflammatory drugs)
* Patients hypersensitive to naproxen sodium or codeine
* Patients who took another analgesic medicine during 24 hours before and/or a nonsteroidal anti-inflammatory medicine during 72 hours before taking study medicine
* Patients with active gastric or duodenum ulcer
* Patients with renal dysfunction and/or a kidney disease
* Patients with severe liver disease
* Patients with rare hereditary galactose intolerance, Lapp lactase insufficiency or glucose-galactose malabsorption problem
* Patients with depression treated by a medicine from monoamine oxidase class
* Patients with uncontrolled hypertension or patients with hypertension that is hardly controlled with medicines
* Patients with a known medical, psychological disturbance or social status that may negatively affect inclusion into the study or patients who may lead to increase in risk for others with inclusion into the study
* Patients with proven clinically important and unstable systemic medical disease
* Patients who have medical contraindication for study medicine
* Patients who are judged by investigator that they will not adhere or adequately adhere to the study protocol
* Patients who participated into another study with another study medicine in the last 4 week
* Patients who intent to donate blood or blood product during the study period or in the following month of the study completion

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Mac Master Questionnaire (WOMAC) | 7 days
Change in Visual Analog Scale (VAS) | 7 days

SECONDARY OUTCOMES:
Change in pain severity in all visits after treatment from baseline (VAS) | 7 days
Functional effects of combination therapy (WOMAC) | 7 days
Change in resting pain after treatment from baseline (WOMAC) | 7 days
Change in activity pain after treatment from baseline (WOMAC) | 7 days
Change in physical function after treatment from baseline (WOMAC) | 7 days
Ratio of rescue medicine use (Rescue medication count) | 7 days
Collection of adverse event reports to evaluate safety of the medicine | 7 days